CLINICAL TRIAL: NCT02805972
Title: Biology and Experience of Eating in Women With Obesity
Acronym: BEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16-19392
Record Dates: First submitted 2016-06-01; First posted 2016-06-20 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Obesity
Keywords: Obesity; Binge eating
MeSH Terms: conditions — Obesity; Bulimia | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naloxone, then Placebo (Experimental): 4 mg / 0.1 ml Naloxone at visit 1, followed by 0.1 ml saline (Placebo) at visit 2 (with a washout period in between the two visits)
  Interventions: Drug: Naloxone; Drug: Placebo
- Placebo, then Naloxone (Experimental): 0.1 ml saline (Placebo) at visit 1, followed by 4 mg / 0.1 ml Naloxone at visit 2 (with a washout period in between the two visits)
  Interventions: Drug: Naloxone; Drug: Placebo

INTERVENTIONS:
Drug: Naloxone — 4 mg / 0.1 ml
  Other Names: Narcan
Drug: Placebo — 0.1 ml
  Other Names: saline

SUMMARY:
The purpose of this study is to understand how the opioid system is involved in eating behavior.

DETAILED DESCRIPTION:
Obesity is associated with greater risk for cardiovascular disease (CVD), stroke, diabetes, and mortality, and is a heterogeneous condition with various causes and thus a diversity of intervention targets. Compulsive overeating afflicts 30% of people seeking obesity treatment and increases risk for CVD factors. This trial involves two participant visits to test whether opioid blockade (Day 1 or 2, depending on randomization), compared to placebo (Day 1 or 2, depending on randomization), will elicit common symptoms of opioid withdrawal, including nausea. Participants will receive each condition on separate days.

ELIGIBILITY:
Inclusion Criteria:

* Obese, as defined by BMI greater than or equal to 30
* Self-reported binge eating as defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), in the last 4 weeks
* If sexually active with men, must agree to use birth control until the final study visit is complete (e.g., barrier methods, oral contraceptive)
* Subject must be able to complete written informed consent procedures and be able to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant or breastfeeding
* Severe hypotension (< 90/60 mmHg)
* Recent or current use of vasoconstrictor or vasodilator medication
* Current or history of diabetes
* Allergies to any ingredients in naloxone hydrochloride
* History of or current alcoholism or drug dependence
* Bulimia Nervosa as defined in DSM 5
* Current or past use of opiate-containing medications in the last 30 days
* Plan to use opiate-containing medications during study participation period
* Medical conditions that are contraindicated with intranasal procedures: Nasal septal abnormalities, nasal trauma, epistaxis, excessive nasal mucus, and intranasal damage caused by the use of substances (e.g., cocaine)
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Naloxone, Then Placebo: At the first intervention visit, participants were administered Naloxone, 4 mg / 0.1 ml, intranasally, after eating. After the washout period, at the second intervention visit, participants were administered the Placebo (saline), 0.1 ml, intranasally, after eating.
- Experimental: Placebo, Then Naloxone: At the first intervention visit, participants were administered the Placebo (saline), 0.1 ml, intranasally, after eating. After the washout period, at the second intervention visit, participants were administered Naloxone, 4 mg / 0.1 ml, intranasally, after eating.
Period: Intervention Visit 1
Arm/Group | Experimental: Naloxone, Then Placebo | Experimental: Placebo, Then Naloxone
Started | 23 | 18
Completed | 23 | 18
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Experimental: Naloxone, Then Placebo | Experimental: Placebo, Then Naloxone
Started | 23 | 18
Completed | 20 | 18
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0
Period: Intervention Visit 2
Arm/Group | Experimental: Naloxone, Then Placebo | Experimental: Placebo, Then Naloxone
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Naloxone, Then Placebo: At visit 1, participants were administered Naloxone, 4 mg/ 0.1 ml, intranasally, after eating. After the washout period between visits, at visit 2, participants were administered the Placebo (saline), 0.1 ml, intranasally, after eating.
- Placebo, Then Naloxone: At visit 1, participants were administered the Placebo (saline), 0.1 ml, intranasally, after eating. After the washout period between visits, at visit 2, participants were administered Naloxone, 4 mg/ 0.1 ml, intranasally, after eating.
- Total: Total of all reporting groups
Arm/Group | Naloxone, Then Placebo | Placebo, Then Naloxone | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 18 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.5) | 33.1 (6.5) | 31.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 23 | 15 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 2
  Asian or Pacific Islander | 3 | 0 | 3
  White | 16 | 15 | 31
  More than one race | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 18 | 41
Weight, kg [Mean (Standard Deviation); unit: kilograms] — Participants were weighted two times at baseline and the average of two measures was used (weight in kilograms).
  kilograms | 104.3 (23.9) | 99.5 (17.0) | 102.2 (21.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) was calculated from the mean of duplicate weight measurements, and the height measurement, at baseline. BMI units are kilograms per meter squared (kg/m^2)
  kg/m^2 | 38.1 (7.1) | 36.4 (4.2) | 37.3 (6.0)
Impulsivity [Mean (Standard Deviation); unit: Probability] — Impulsivity, measured by the Delayed Discounting cognitive task, based on a series of 30 computer-administered trials or questions. Indifference points (a measure of how much a person values a delayed reward) are determined for time delays of: 1 day, 7 days, 30 days, 180 days, and 365 days, and these are used to calculate an Area Under the Curve which ranges from 0 to 1 (lower numbers indicate higher impulsivity) as a metric of probability.
  Probability | 0.69 (0.21) | 0.57 (0.29) | 0.64 (0.25)
Reward-driven Eating (RED) scale [Mean (Standard Deviation); unit: units on a scale] — Total score ranges from 0 (lower reward-driven eating) to 52 (higher reward-driven eating).
  units on a scale | 38.1 (6.1) | 36.8 (5.2) | 37.5 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Nausea at 10 Minutes Post Treatment
Description: Dichotomized response on the "I feel nauseous" question of the Subjective Opiate Withdrawal Scale, at 10 minutes after the listed intervention (among participants who completed both intervention visits). Response 0 = absence of nausea, 1 = presence of nausea.
Time Frame: 10 minutes post-treatment
Population: All participants who received Naloxone, then Placebo, or Placebo, then Naloxone, by participating in both study intervention visits.
Measure: Count of Participants; unit: Participants
Groups:
- Naloxone: 4 mg / 0.1 ml naloxone
  Naloxone: 4 mg / 0.1 ml
- Placebo: 0.1 ml saline
  Placebo: 0.1 ml
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
Participants | 17 | 18

2. Primary Outcome: Number of Participants Who Reported Nausea at 30 Minutes Post Treatment
Description: Dichotomized response on the "I feel nauseous" question of the Subjective Opiate Withdrawal Scale, at 30 minutes after the listed intervention (among participants who completed both intervention visits). Response 0 = absence of nausea, 1 = presence of nausea.
Time Frame: 30 minutes post-treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
Participants | 13 | 11

3. Secondary Outcome: Cortisol
Description: Geometric Mean Salivary Cortisol level.
Time Frame: 25 minutes post-treatment
Population: Participants 25 minutes after Naloxone or Placebo administration, among those who completed both intervention visits
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Groups:
- Naloxone: Measurement of Cortisol here reported 25 min post Naloxone, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
- Placebo: Measurement of Cortisol here reported 25 min post Placebo, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
nmol/L | 3.22 (2.18) | 3.37 (1.96)

4. Secondary Outcome: Cortisol
Description: Geometric Mean Salivary Cortisol level.
Time Frame: 55 minutes post-treatment
Population: Participants 55 minutes after Naloxone or Placebo administration, among those who completed both intervention visits
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Groups:
- Naloxone: Measurement of Cortisol here reported 55 min post Naloxone, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
- Placebo: Measurement of Cortisol here reported 55 min post Placebo, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
nmol/L | 3.61 (2.26) | 2.90 (2.19)
Statistical Analysis 1: Comparison: Naloxone; We compared cortisol values at 55 minutes, within person, across conditions. We Winsorized one participant's values for the placebo visit where values were between 2-4x above the 99th percentile value in the data and then log-transformed the data; Test type: Superiority — The null hypothesis is that there would be no difference across the Naloxone and placebo conditions. The alternative hypothesis is that the cortisol value would be higher in the Naloxone condition than in the placebo condition; p = .067, t-test, 2 sided — If the Winsorized value is excluded from analyses altogether, the P value is .012; Cortisol was log transformed for the statistical test, and the reported mean difference was exponentiated back to the original units of nmol/L below; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [0.98 to 1.61]

5. Secondary Outcome: Subjective Opiate Withdrawal Scale
Description: Summed score of Subjective Opiate Withdrawal Scale (SOWS). Scale consists of 16 items answered on a 5 point numeric rating scale. Score range is 0 (lesser withdrawal symptoms) to 64 (greater withdrawal symptoms). Scores were assessed at 10 minutes after Naloxone, and at a separate visit, 10 minutes after Placebo, among participants who completed both study visits.
Time Frame: 10 minutes post-treatment
Population: Measurement of Subjective Opiate Withdrawal Scale here reported 10 min post Naloxone or 10 minutes after Placebo, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Naloxone: Measurement of SOWS after Naloxone, among all participants who received Naloxone: 4 mg / 0.1 ml post eating at visit 1 and after a washout period, Placebo (saline): 0.1 ml post eating at visit 2, or were randomized to instead receive the same dosage of Placebo at visit 1 followed by a washout period and then Naloxone at visit 2.
- Placebo: Measurement of SOWS after Placebo, among all participants who received Naloxone: 4 mg / 0.1 ml post eating at visit 1 and after a washout period, Placebo (saline): 0.1 ml post eating at visit 2, or were randomized to instead receive the same dosage of Placebo at visit 1 followed by a washout period and then Naloxone at visit 2.
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale | 5.67 (3.65) | 5.03 (3.58)

6. Secondary Outcome: Subjective Opiate Withdrawal Scale (Abbreviated)
Description: Mean score on subset of 5 items (which used a 5 point numeric rating response scale) from the Subjective Opiate Withdrawal Scale (SOWS). This summed score can range from 0 (corresponding to lesser withdrawal symptoms) to 20 (corresponding to greater withdrawal symptoms).
Time Frame: 30 minutes post-treatment
Population: Measurement of the abbreviated SOWS here reported 30 min post Naloxone or 30 min post Placebo, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Naloxone: Measurement of the abbreviated Subjective Opiate Withdrawal Scale here reported 30 min post Naloxone, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
- Placebo: Measurement of the abbreviated Subjective Opiate Withdrawal Scale here reported 30 min post Placebo, among all participants who received Naloxone (4mg / 0.1 ml), then after a washout period, received Placebo (saline, 0.1 ml), or Placebo, then after a washout period, received Naloxone, by participating in both study intervention visits.
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale | 1.42 (1.35) | 1.53 (1.50)

7. Other Pre Specified Outcome: Reward-Driven Eating Scale (RED)
Description: Reward-Driven Eating Scale (RED) total score ranges from 0 (lower reward-driven eating) to 52 (higher reward-driven eating).
Time Frame: Evaluated before study visit 1
Population: All eligible participants who were randomized to either order of intervention conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Naloxone, Then Placebo: Includes all participants randomized to receive Naloxone (4mg / 0.1 ml), then after a washout period, receive Placebo (saline, 0.1 ml), with reward-driven eating evaluated before the first study intervention.
- Placebo, Then Naloxone: Includes all participants randomized to receive Placebo (saline, 0.1 ml), then after a washout period, receive Naloxone (4mg / 0.1 ml), with reward-driven eating evaluated before the first study intervention.
Arm/Group | Experimental: Naloxone, Then Placebo | Placebo, Then Naloxone
Number analyzed (Participants) | 23 | 18
score on a scale | 38.1 (6.1) | 36.8 (5.2)

8. Other Pre Specified Outcome: Impulsivity (Delayed Discounting)
Description: Impulsivity, measured by the Delayed Discounting cognitive task, based on a series of 30 computer-administered trials or questions. Indifference points (a measure of how much a person values a delayed reward) are determined for time delays of: 1 day, 7 days, 30 days, 180 days, and 365 days, and these are used to calculate an Area Under the Curve which ranges from 0 to 1 (lower numbers indicate higher impulsivity) as a metric of probability.
Time Frame: Impulsivity was assessed before the study visit 1 intervention.
Population: All eligible participants randomized to either order of the intervention.
Measure: Mean (Standard Deviation); unit: Probability
Arm/Group | Experimental: Naloxone, Then Placebo | Placebo, Then Naloxone
Number analyzed (Participants) | 23 | 18
Probability | 0.69 (0.21) | 0.57 (0.29)

ADVERSE EVENTS:
Time Frame: Two days (each study intervention visit was conducted over approximately 4 hours, with the 2 interventions administered on a total of 2 separate visit days).
Description: The definition used did not differ from that of clinicaltrials.gov
Groups:
- Naloxone, Then Placebo: Visit 1 intervention condition: 4 mg / 0.1 ml Naloxone, followed by visit 2 condition: 0.1 ml Placebo (saline)
- Placebo, Then Naloxone: Visit 1 intervention condition: 0.1 ml Placebo (saline), followed by visit 2 condition: 4 mg / 0.1 ml Naloxone
Arm/Group | Naloxone, Then Placebo | Placebo, Then Naloxone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/18
Other Adverse Events (participants affected / at risk) | 0/23 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT02805972/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT02805972/ICF_001.pdf